CLINICAL TRIAL: NCT00683020
Title: Harnessing Health IT for Self-Management Support and Medication Activation in a Medicaid Health Plan
Acronym: SMARTSteps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco Health Plan (SFHP) (Unknown); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R18HS017261 (AHRQ)
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Results first posted 2013-05-15 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Diabetes
Keywords: Chronic Diseases; Diabetes; Vulnerable population; Urban populations; Disease Management; Health Information Technology; Safety; Health Literacy; Level of English Proficiency
MeSH Terms: conditions — Diabetes Mellitus; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ATSM Intervention (Active Comparator): ATSM Intervention: Automated Telephone Self-Management Support.
  Interventions: Behavioral: ATSM Intervention
- WAIT LIST Control (No Intervention): WAIT LIST Control: six month Wait List.

INTERVENTIONS:
Behavioral: ATSM Intervention — The ATSM system is designed to promote the efficiency of a care manager by having her focus outreach phone calls to patients who, by virtue of their responses to the ATSM system, report a need for further support. The purpose of these call-backs is to have the care manager directly engage patients in setting goals and developing an action plan to improve their overall health. The care manager is trained to perform motivational interviewing, assess and overcome barriers to health communication.
  For some patients, the ATSM system as described above is augmented by additional phone communications from care manager to patient, triggered by health IT derived from 2 additional data sources: SFHP pharmacy claims data and CHNSF diabetes registry. The latter combines clinical data (labs and blood pressure). Based on clinical criteria, the ATSM system will alert care manager to make additional calls to patients.
  Other Names: ATSM: Automated Telephone Self-Management Support
  Arms: ATSM Intervention

SUMMARY:
To measure the effects of a Medical health plan-directed automated telephone self-management support system (ATSM) on patient outcomes among ethnically diverse health plan enrollees with diabetes.

DETAILED DESCRIPTION:
We will be conducting an evaluation of a quality improvement initiative that the San Francisco Health Plan (SFHP), a large Medicaid managed care plan in SF, is conducting for approximately 500 SFHP enrollees with diabetes who are attending 4 Community Health Network Clinics in San Francisco (CHNSF) over a two year period. The intervention that SFHP is implementing is Automated Telephone Support Management (ATSM), a health IT innovation used as adjunct to care management. The partnership with University of California, San Francisco-San Francisco General Hospital (UCSF-SFGH) researchers is based on previous work we have done in the CHNSF regarding using ATSM among diabetes patients to improve self-management activities and other health outcomes,but in the current demonstration project and evaluation, the recruitment of participants and implementation of the intervention will be done by the SFHP; UCSF will only conduct an evaluation. The Governing Board at the SFHP decided to adopt the ATSM model for its growing number of diabetes patients, to dedicate nursing staff to respond to ATSM data and engage with enrollees and their providers, to underwrite the costs of ATSM implementation, to randomly assign their patients to one of two types of ATSM (one that involves medication review/intensification vs. one that only delivers behavioral support), and to contact eligible SFHP members for ATSM and also to briefly describe the evaluation study to be carried out by UCSF. We, as UCSF researchers, will evaluate the impact of the interventions on patient outcomes. There will be limited contact with patients by the UCSF research team. UCSF research staff will only contact patients after SFHP has determined that their patients are interested in being contacted about the evaluation; and there will be no collection of personal health information by UCSF evaluators. UCSF research staff will conduct a telephone survey after verbal consent procedures, at baseline and 6 months (and for patients wait-listed, again at 12 months), for patients participating in the ATSM intervention. The SFHP will maintain an identification (ID) link between patients who are in the intervention and who are conducted about the evaluation, but they will not have patient-linked survey data, nor will UCSF have linked health-related data from the SFHP regarding patient outcomes, although de-identified data will be included in the UCSF evaluation. UCSF will conduct the quantitative data analyses of de-identified data provided to us by the SFHP at set times over the study period to examine the impact of the interventions on clinical outcomes. The evaluation will focus on the effects of ATSM on both patient-centered outcomes and on clinical outcomes through this "real-world" effectiveness study. The fact that recruitment and implementation will be carried out by SFHP, that SFHP will maintain the link to patients in the evaluation but will not have the survey data linked to individuals, and that only SFHP will have control over the personal health information of patients, has important implications for generalizability.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes diagnosis
* Attend one of 4 CHNSF clinics
* Ages 18 or above
* Speak English, Spanish or Cantonese
* Have a touch tone phone
* Have had one or more clinic visits in the preceding 24 months
* Will be in the SF Bay Area for the following six months

Exclusion Criteria:

* Pregnant
* Unable to provide verbal consent
* Leaving the region in the next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2009-04; Primary Completion 2011-11 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dean Schillinger, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Center for Vulnerable Populations, San Francisco, California, United States

REFERENCES:
- [Derived] Ratanawongsa N, Quan J, Handley MA, Sarkar U, Schillinger D. Language-concordant automated telephone queries to assess medication adherence in a diverse population: a cross-sectional analysis of convergent validity with pharmacy claims. BMC Health Serv Res. 2018 Apr 6;18(1):254. doi: 10.1186/s12913-018-3071-4. PMID 29625571
- [Derived] Quan J, Lee AK, Handley MA, Ratanawongsa N, Sarkar U, Tseng S, Schillinger D. Automated Telephone Self-Management Support for Diabetes in a Low-Income Health Plan: A Health Care Utilization and Cost Analysis. Popul Health Manag. 2015 Dec;18(6):412-20. doi: 10.1089/pop.2014.0154. Epub 2015 Jun 23. PMID 26102298
- [Derived] Ratanawongsa N, Handley MA, Quan J, Sarkar U, Pfeifer K, Soria C, Schillinger D. Quasi-experimental trial of diabetes Self-Management Automated and Real-Time Telephonic Support (SMARTSteps) in a Medicaid managed care plan: study protocol. BMC Health Serv Res. 2012 Jan 26;12:22. doi: 10.1186/1472-6963-12-22. PMID 22280514

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study sample was drawn from San Francisco Health Plan The study sample was drawn April 2009 - March 2011 from San Francisco Health Plan (SFHP) members who received primary care at one of four publicly-funded clinics in the Community Health Network of San Francisco (CHNSF).
Pre-assignment Details: SFHP members deemed eligible were English-, Cantonese-, or Spanish-speaking adults (age 18 or above) with ≥1 primary care clinic visit in the preceding 24 months, had diabetes diagnosis, and access to a touch-tone phone. Members who were pregnant, unable to provide verbal consent, or leaving the region in the next 12 months were ineligible.
Period: Overall Study
Arm/Group | ATSM Intervention | WAIT LIST Control
Started | 182 | 180
Completed | 127 | 125
Not Completed | 55 | 55

BASELINE CHARACTERISTICS:
Population: Data is based on the 252 participants with both baseline and 6-month follow-up measures.
Groups:
- Total: Total of all reporting groups
Arm/Group | ATSM Intervention | WAIT LIST Control | Total
Number analyzed (Participants) | 127 | 125 | 252
Age Continuous [Mean (Standard Deviation); unit: years] | 56.5 (7.9) | 55.0 (8.6) | 55.7 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 89 | 187
  Male | 29 | 36 | 65
Race/Ethnicity, Customized [Number; unit: Participants]
  Latino | 32 | 25 | 57
  Black / African-American | 7 | 12 | 19
  Asian / Pacific Islander | 77 | 78 | 155
  White / Caucasian | 7 | 9 | 16
  Multi-Ethnic / Other | 4 | 1 | 5
Birth Place [Number; unit: Participants]
  Outside U.S. | 110 | 106 | 216
  Inside U.S. | 17 | 19 | 36
Language [Number; unit: Participants]
  Cantonese | 69 | 69 | 138
  Spanish | 25 | 23 | 48
  English | 33 | 33 | 66
Language Concordance with Primary Care Provider [Number; unit: Participants] — Data is based on the 252 participants with baseline and 6-month follow-up measures, Cantonese- or Spanish-speaking, and with a regular primary care provider.
  Participants
    Concordant | 33 | 26 | 59
    Discordant | 57 | 62 | 119
Educational Attainment [Number; unit: Participants]
  8th grade education or less | 50 | 58 | 108
  Some high school | 13 | 12 | 25
  High school graduate or GED | 33 | 22 | 55
  College graduate or above | 31 | 33 | 64
Health Literacy [Number; unit: Participants] — Data is based on the 252 participants with both baseline and 6-month follow-up measures and with answers to all health literacy questions.
  Participants
    Limited | 58 | 50 | 108
    Adequate | 68 | 75 | 143
Employment Status [Number; unit: Participants]
  Employed full-time | 28 | 26 | 54
  Part-time | 63 | 58 | 121
  Unemployed | 12 | 15 | 27
  Disabled | 7 | 13 | 20
  Homemaker / Retired / Other | 17 | 13 | 30
Annual Household Income [Number; unit: Participants] — Data is based on the 252 participants with both baseline and 6-month follow-up measures and with answer to the question on annual household income.
  Participants
    ≤ $20,000 | 73 | 75 | 148
    $20,001 - $30,000 | 24 | 25 | 49
    >$30,000 | 19 | 19 | 38
Financial Class - Insurance Type [Number; unit: Participants] — Data is based on the 252 participants with both baseline and 6-month follow-up measures and with financial class information.
  Participants
    Medicaid | 28 | 22 | 50
    Medicare | 4 | 7 | 11
    Uninsured / Commercial | 1 | 2 | 3
    Healthy Worker / Healthy San Francisco | 93 | 94 | 187
Diabetes Duration [Mean (Standard Deviation); unit: Years] | 6.9 (5.9) | 7.2 (5.4) | 7.0 (5.7)
Insulin Treatment [Number; unit: Participants]
  Yes | 25 | 18 | 43
  No | 102 | 107 | 209
Hemoglobin A1c [Number; unit: Participants] — Data is based on the 252 participants with both baseline and 6-month follow-up measures and with Hemoglobin A1c data.
  Participants
    > 8.0% | 37 | 29 | 66
    ≤ 8.0% | 87 | 90 | 177
Hemoglobin A1c [Mean (Standard Deviation); unit: %] — Data is based on the 252 participants with both baseline and 6-month follow-up measures and with Hemoglobin A1c data.
  % | 7.8 (1.6) | 7.5 (1.3) | 7.7 (1.5)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 127.3 (17.3) | 128.1 (18.2) | 127.7 (17.7)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 72.9 (9.3) | 76.1 (9.9) | 74.5 (9.7)
Low-density Lipoprotein [Mean (Standard Deviation); unit: mg/dL] | 92.7 (30.3) | 93.5 (31.5) | 93.1 (30.8)

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Physical Component Summary of the SF-12 Health Survey
Description: The SF-12 Health Survey (SF-12) is a 12-item short-form survey used to measure health status and monitor health outcomes. The survey asks about various health aspects, including physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health (psychological distress and psychological well-being). Two summary measures are derived: the Physical and the Mental Health Component Summary. For each component summary, survey items were weighted and summed to create a summary score between 0 and 100 with higher score indicating better functioning and outcome. Change is calculated as 6-month score minus baseline score.
Time Frame: Baseline and 6 months
Population: The Participant Flow Module numbers are the numbers of participants in the particular categories of the module. However, the number of participants analyzed counts only those participants who have both baseline and 6-month follow-up outcome data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ATSM Intervention | WAIT LIST Control
Number analyzed (Participants) | 119 | 119
units on a scale | 1.3 (0.7) | -0.7 (0.7)
Statistical Analysis 1: Comparison: ATSM Intervention vs WAIT LIST Control; Test type: Non-Inferiority or Equivalence — Mean changes in comparison groups are not equal; p = 0.03, Regression, Linear; Adjusted for baseline values; Mean Difference (Net) = 2.0, 95% CI 2-sided [0.1 to 3.9], Standard Error of Mean 0.9

2. Primary Outcome: Changes in the Mental Component Summary of the SF-12 Health Survey
Description: as for outcome 1
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ATSM Intervention | WAIT LIST Control
Number analyzed (Participants) | 119 | 119
units on a scale | 1.4 (0.8) | 0.0 (0.8)
Statistical Analysis 1: Comparison: ATSM Intervention vs WAIT LIST Control; Test type: Non-Inferiority or Equivalence — Mean changes in comparison groups are not equal; p = 0.23, Regression, Linear; Adjusted for baseline values; Mean Difference (Net) = 1.4, 95% CI 2-sided [-0.9 to 3.6], Standard Error of Mean 1.2

3. Secondary Outcome: Number of Days Spent in Bed Due to Illness
Description: A measure of patients' functional status is ascertained by asking patients the following question: "In the last 30 days, how many days did health problems keep you in bed for all or most of the day?" Number of days may range from 0 to 30, with lower number of days indicating better functional status. Because a negative binomial model was used to analyze the data for number of days spent in bed due to illness, log means are reported. A log mean is the natural (base e) logarithm of the mean (in this context specifically, the mean number of days spent in bed due to illness). To calculate the mean, one raises e by the number given as the log mean. Lower log means indicate better functional status.
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: log days
Arm/Group | ATSM Intervention | WAIT LIST Control
Number analyzed (Participants) | 127 | 124
log days | 0.02 (0.3) [0.010 to 0.03] | 0.03 (0.3) [0.016 to 0.051]
Statistical Analysis 1: Comparison: ATSM Intervention vs WAIT LIST Control; Test type: Non-Inferiority or Equivalence — Days in comparison groups are not equal; p = 0.25, Negative Binomial Models; Adjusted for baseline values; Rate Ratio = 0.6, 95% CI 2-sided [0.3 to 1.4]

4. Secondary Outcome: Proportion of Patients Reporting Diabetes Interference of Normal Daily Activities
Description: A measure of diabetes interference on patients is ascertained by asking patients the following question: "In the last 6 months, how often has your diabetes kept you from doing your normal daily activities, such as going to work, grocery shopping, and taking care of yourself and others?" Responses consist of 6 possible options: "Always", "Almost Always", "Often", "Sometimes", "Almost Never", and "Never". These responses are grouped into 2 categories, with one category consisting of "Always", "Almost Always", and "Often" responses while the other category consists of the remaining responses. The proportion of patients reporting diabetes interference is the number of patients in the first category divided by the number of patients in the 2 categories combined.
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: proportion of patients
Arm/Group | ATSM Intervention | WAIT LIST Control
Number analyzed (Participants) | 127 | 124
proportion of patients | 0.039 [0.1 to 0.6] | 0.088 [0.0 to 0.0]
Statistical Analysis 1: Comparison: ATSM Intervention vs WAIT LIST Control; Test type: Non-Inferiority or Equivalence — Proportions in comparison groups are not equal; p = 0.18, Regression, Logistic; Adjusted for baseline values; Odds Ratio (OR) = 0.5, 95% CI 2-sided [0.2 to 1.4]

5. Secondary Outcome: Changes in Diabetes Self-management Behaviors as Measured by Summary of Diabetes Self-Care Activities (SDSCA) Scale
Description: The Summary of Diabetes Self-Care Activities (SDSCA) Measure is a brief self-report questionnaire on diabetes self-management behaviors. The questionnaire assesses the frequency with which a patient followed a diabetes routine over the prior 7 days in five domains: diet, exercise, blood-glucose testing, foot care, and medication adherence. Based on SDSCA measure's author's recommendations, two separate scores are derived: a Diabetes Self-management Behaviors score and a Self-reported Medication Adherence score. For the Diabetes Self-management Behaviors score, all items pertaining to diet, exercise, blood glucose testing, and foot care are averaged. For the Self-reported Medication Adherence score, all items pertaining to medication use are averaged. For both scores, the result is an average score between 0 and 7 with higher score indicating better diabetes self-management behavior or better medication adherence. Change is calculated as 6-month score minus baseline score.
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ATSM Intervention | WAIT LIST Control
Number analyzed (Participants) | 127 | 125
units on a scale | 0.7 (0.4) | 0.08 (0.08)
Statistical Analysis 1: Comparison: ATSM Intervention vs WAIT LIST Control; Test type: Non-Inferiority or Equivalence — Mean changes in comparison groups are not equal; p = 0.008, Regression, Linear; Adjusted for baseline values; Mean Difference (Net) = 0.3, 95% CI 2-sided [0.1 to 0.5], Standard Error of Mean 0.1

6. Secondary Outcome: Changes in Self-reported Medication Adherence as Measured by Summary of Diabetes Self-Care Activities (SDSCA) Scale
Description: as for outcome 5
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ATSM Intervention | WAIT LIST Control
Number analyzed (Participants) | 122 | 117
units on a scale | 0.2 (0.06) | 0.2 (0.06)
Statistical Analysis 1: Comparison: ATSM Intervention vs WAIT LIST Control; Test type: Non-Inferiority or Equivalence — Mean changes in comparison groups are not equal; p = 0.87, Regression, Linear; Adjusted for baseline values; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.2 to 0.2], Standard Error of Mean 0.1

7. Secondary Outcome: Changes in Diabetes Self-efficacy as Measured by Diabetes Quality Improvement Project's Patient Self-Management Scale
Description: The Patient Self-Management Scale was derived from a questionnaire used in the Diabetes Quality Improvement Project. The scale is designed to reflect patients' assessment of their ability to manage aspects of diabetes self-care in 5 separate areas (medication, diet, exercise, blood glucose monitoring, and foot care). Respondents are asked how difficult over the past 6 months has it been to follow exactly as their doctor who takes care of their diabetes suggested. Possible scores for each scale item range from 0 to 100 with higher score indicating more self-efficacy. Total scale score is calculated as the average across all items. Change is calculated as 6-month score minus baseline score.
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ATSM Intervention | WAIT LIST Control
Number analyzed (Participants) | 127 | 125
units on a scale | 6.8 (1.1) | 5.7 (1.1)
Statistical Analysis 1: Comparison: ATSM Intervention vs WAIT LIST Control; Test type: Non-Inferiority or Equivalence — Mean changes in comparison groups are not equal; p = 0.49, Regression, Linear; Adjusted for baseline values; Mean Difference (Net) = 1.1, 95% CI 2-sided [-2.1 to 4.2], Standard Error of Mean 1.6

8. Secondary Outcome: Changes in Patient-centeredness of Care as Measured by Patient Assessment of Chronic Illness Care (PACIC) Scale
Description: The Patient Assessment of Chronic Illness Care (PACIC) is a 20-item patient report instrument that measures patients' perspectives on the structure of their care and collects patient reports on the extent to which they have received specific clinical services and actions during the past 6 months that are aligned with the Chronic Care Model. The scale is intended to assess the receipt of care that is patient-centered, proactive, planned and includes collaborative goal setting, problem-solving and follow-up support. Each instrument item is scored on a 5-point scale ranging from 1 to 5 with higher score indicating better care. Scores are transformed to a 100-point scale (0-100) and averaged across all items to create a total scale score. Higher transformed and total scale scores indicate better care. Change is calculated as 6-month score minus baseline score.
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ATSM Intervention | WAIT LIST Control
Number analyzed (Participants) | 127 | 125
units on a scale | 11.3 (1.5) | 10.0 (1.6)
Statistical Analysis 1: Comparison: ATSM Intervention vs WAIT LIST Control; Test type: Non-Inferiority or Equivalence — Mean changes in comparison groups are not equal; p = 0.54, Regression, Linear; Adjusted for baseline values; Mean Difference (Net) = 1.3, 95% CI 2-sided [-3.0 to 5.6], Standard Error of Mean 2.2

9. Secondary Outcome: Changes in Patient-centeredness of Care as Measured by Interpersonal Processes of Care (IPC) Scale
Description: The Interpersonal Processes of Care (IPC) is an 18-item patient report instrument that measures patients' perspectives on the structure of their care and collects patient reports on providers' communication over the prior 6 months. The scale is intended to measure patients' assessment of providers' communication within 3 broad domains: communication (e.g., lack of clarity), decision making (e.g., patient-centered decision making), and interpersonal style (e.g., friendliness). Each instrument item is scored on a 5-point scale ranging from 1 to 5. Scores are transformed to a 100-point scale and averaged across all items to create a total scale score. Higher total scores indicate better communication. Change is calculated as 6-month score minus baseline score.
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ATSM Intervention | WAIT LIST Control
Number analyzed (Participants) | 127 | 125
units on a scale | -1.8 (0.9) | -3.8 (0.9)
Statistical Analysis 1: Comparison: ATSM Intervention vs WAIT LIST Control; Test type: Non-Inferiority or Equivalence — Mean changes in comparison groups are not equal; p = 0.11, Regression, Linear; Adjusted for baseline values; Mean Difference (Net) = 2.0, 95% CI 2-sided [-0.4 to 4.4], Standard Error of Mean 1.2

10. Secondary Outcome: Changes in Hemoglobin A1c Levels
Description: Hemoglobin A1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. As the average amount of plasma glucose increases, the fraction of hemoglobin A1c increases in a predictable way. This serves as a marker for average blood glucose levels over the previous months prior to the measurement. Higher amounts of hemoglobin A1c indicate poorer control of blood glucose levels and have been associated with cardiovascular disease. Change is calculated as 6-month level minus baseline level.
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | ATSM Intervention | WAIT LIST Control
Number analyzed (Participants) | 56 | 50
percentage | -0.5 (0.1) | -0.2 (0.1)
Statistical Analysis 1: Comparison: ATSM Intervention vs WAIT LIST Control; Test type: Non-Inferiority or Equivalence — Mean changes in comparison groups are not equal; p = 0.13, Regression, Linear; Adjusted for baseline values; Mean Difference (Net) = -0.3, 95% CI 2-sided [-0.6 to 0.1], Standard Error of Mean 0.2

11. Secondary Outcome: Changes in Systolic Blood Pressure (SBP)
Description: Systolic blood pressure is the pressure exerted on arteries and vessels by the heart when it contracts and pushes blood through the arteries to the rest of the body. Change is calculated as 6-month pressure minus baseline pressure.
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | ATSM Intervention | WAIT LIST Control
Number analyzed (Participants) | 79 | 88
mm Hg | 0.2 (1.7) | -0.4 (1.6)
Statistical Analysis 1: Comparison: ATSM Intervention vs WAIT LIST Control; Test type: Non-Inferiority or Equivalence — Mean changes in comparison groups are not equal; p = 0.78, Regression, Linear; Adjusted for baseline values; Mean Difference (Net) = 0.6, 95% CI 2-sided [-3.8 to 5.1], Standard Error of Mean 2.3

12. Secondary Outcome: Changes in Diastolic Blood Pressure (DBP)
Description: Diastolic blood pressure is the pressure exerted on the walls of the arteries and vessels in between heart beats, when the heart is relaxed and dilated, filling with blood. Change is calculated as 6-month pressure minus baseline pressure.
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | ATSM Intervention | WAIT LIST Control
Number analyzed (Participants) | 79 | 88
mm Hg | 1.2 (1.0) | -0.9 (1.0)
Statistical Analysis 1: Comparison: ATSM Intervention vs WAIT LIST Control; Test type: Non-Inferiority or Equivalence — Mean changes in comparison groups are not equal; p = 0.13, Regression, Linear; Adjusted for baseline values; Mean Difference (Net) = 2.1, 95% CI 2-sided [-0.6 to 4.9], Standard Error of Mean 1.4

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | ATSM Intervention | WAIT LIST Control
Serious Adverse Events (participants affected / at risk) | 0/182 | 0/180
Other Adverse Events (participants affected / at risk) | 0/182 | 0/180

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes